CLINICAL TRIAL: NCT04648267
Title: Factors Affecting Split Thickness Skin Graft Success Rates in Patients Who Underwent a Radial Forearm or Fibula Free Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Neils Kokot, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-20-00490
Record Dates: First submitted 2020-11-14; First posted 2020-12-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Skin Graft Complications
Keywords: Split thickness skin graft; radial forearm free flap; fibula free flap
MeSH Terms: interventions — POLR1G protein, human; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigators evaluating the skin grafts with adobe photoshop will be masked and will not know which skin graft belonged to which patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients who have the cast and bolster on for standard 5 days after their radial forearm free flap and 7 days after their fibula free falp
  Interventions: Other: Standard of care
- Experimental group (Experimental): Patients who have the cast and bolster on for 10-14 days
  Interventions: Other: Cast and bolster placement duration

INTERVENTIONS:
Other: Cast and bolster placement duration — The intervention is increasing the duration of cast and bolster placement on split thickness skin graft sites.
  Arms: Experimental group
Other: Standard of care — This will be standard of care - the patient will have his cast and bolster on for 5-7 days
  Arms: Control group

SUMMARY:
Fibula free flaps (FFF) and radial forearm free flaps (RFFF) are necessary to reconstruct parts of the face after cancer surgery, traumas, or debilitating infections. Oftentimes, after we take the flap from the arm or leg, there is a large skin defect that must be filled. A split thickness skin graft (STSG) usually from the thigh can be used to fill this defect. Split thickness skin grafts get their blood supply from the underlying tissue, Hence, pressure must be applied to the skin grafts to ensure that they "stick" to the underlying tissue and are properly perfused. A bolster and cast is placed onto the skin graft to apply pressure and to immobilize the skin graft to optimize healing. However, skin grafts still often do not take well. Thus, the objective of this study is to see if the duration of the cast and bolster over the skin graft has an effect on how well it integrates into the wound bed.

The study will compare 2 groups: the standard of care 5-7 day cast group versus the experiment 10-14 day cast group. The hypothesis is that people with longer cast and bolster duration will have better healing rates. Surveys will also be administered to see if cast and bolster duration will affect quality of life and self-esteem.

DETAILED DESCRIPTION:
This will be a prospective randomized control trial with a recruitment goal of 220 patients. One hundred and ten (110) patients will have undergone a split thickness skin graft (STSG) to reconstruct the fibula free flap (FFF) donor site and another one hundred and ten (110) patients will be for those with a radial forearm free flap (RFFF) donor site. This is anticipated to be a 5 year study.

Patients will be recruited in clinic. The study will be discussed at their pre-surgery evaluation visit and patients will be provided with a copy of the consent form to take home to discuss whether or not they wish to proceed with the study. On the day of the surgery, should the patients decide on joining the study, they will be consented and asked to fill out pre-surgery surveys. These surveys are the quality of life 36 item short form survey (SF 36) and a Rosenberg self-esteem survey.

Participants will be randomized to either the standard or the experimental group and this information will be placed in an opaque envelope attached to the consent. Participants then undergo surgery and receive routine post-operative care as per standard of care. After surgery on post operative day 1, one of the co-investigators will open the envelope which will reveal whether the participant is to have the cast and bolster for 5-7 days or 10-14 days. Participants who have their casts and bolsters on for 5-7 days will have them removed before discharge and those who are assigned to the longer group will have them taken off in clinic at their first post-operative visit.

At their one month follow up appointment, a picture will be taken of the donor site. Participants will also be asked to fill out a quality of life 36 item short form survey (SF 36) and a Rosenberg self-esteem survey directly on Redcap. Participants do not have to make extra trips to the physician's office. These pictures and surveys will be administered at their routine office visits. At 3 month, the participant will receive the same surveys again by mail or email, per their preference. Once they have completed these surveys at 3 months, they will have completed their portion of the study.

The investigators will then analyze the skin graft pictures on Adobe Photoshop. All of the photos of the grafts will be de-identified and the people analyzing the pictures will be blinded. They will estimate the percentage of the graft that has healed well or "take"

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent a radial forearm free flap or fibula free flap and split thickness skin graft placed over the donor site

Exclusion Criteria:

* Patients who cannot make informed decisions
* Patients who cannot make their one month post-operative appointment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
The effect of cast and bolster duration on split thickness skin graft integration | The patient will be assessed one month after surgery to take a picture of their skin grafts.
  At one month, we will take pictures in clinic of the split thickness skin graft. Afterwards, two blinded investigators will determine how much of the skin graft has integrated. Exposed tendon and muscle indicate that that part of the skin graft has failed. This will be done on Adobe Photoshop and the integration percentage will be scored. The scale will be from 0% to 100%. A higher percentage is a better outcome

SECONDARY OUTCOMES:
The effect of cast duration on self esteem | The surveys will be administered once before surgery, once 1 month after surgery and once 3 months after surgery
  The surveys that will be administered include the Rosenberg self-esteem survey. This is scored on a 4 point Likert scale. A higher score indicates higher self-esteem and a more favorable outcome
The effect of cast duration on quality of life | The surveys will be administered once before surgery, once 1 month after surgery and once 3 months after surgery
  The surveys that will be administered include the Short Form 36 quality of life form (SF 36). It is measured with 8 scales scores. Each scale is then transformed into a percentage from 0 to 100. A higher percentage indicates less disability and a more favorable outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT04648267/Prot_SAP_001.pdf